CLINICAL TRIAL: NCT05522608
Title: Factors Associated With Postoperative Pain in Patients Undergoing Transabdominal Preperitoneal Hernia Repair for Inguinal Hernia
Brief Title: Factors Associated With Postoperative Pain in Patients Undergoing TAPP Hernia Repair for Inguinal Hernia
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Korhan TUNCER, General Surgeon, Tepecik Training and Research Hospital
Other Study IDs: 2021/04-09
Record Dates: First submitted 2022-07-16; First posted 2022-08-31 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Inguinal Hernia; Postoperative Pain
Keywords: inguinal hernia; postoperative pain; transabdominal preperitoneal repair; visual analogue scale
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with postoperative pain: Patients with postoperative pain after transabdominal preperitoneal hernia repair
  Interventions: Procedure: transabdominal preperitoneal hernia repair
- patients without postoperative pain: Patients without postoperative pain after transabdominal preperitoneal hernia repair
  Interventions: Procedure: transabdominal preperitoneal hernia repair

INTERVENTIONS:
Procedure: transabdominal preperitoneal hernia repair — It is made through 3 holes, 10 mm optical port from the umbilicus, and 5 mm ports each from the right and left lower quadrants. The peritoneum is opened a few cm above the defect in the form of an arc. Dissection of the peritoneum, first lateral and then medial to the defect, is performed. It is continued until the pubic bone is found medially and the periphery of the bone is released. The dissection of the cord elements and the sac is completed. Posterior dissection is a very important step to avoid recurrence. Here, the peritoneum is thoroughly dissected posteriorly, the ductus deferens and vessels are removed from the peritoneum so that no recurrence occurs under the patch. 1-2 to the pubic tubercle, 3-5 to the upper edge of the patch, to the upper edge. Staples at the upper edge should remain above the iliopubic tract, no staples should be placed below. The patch is closed by overlapping the peritoneal leaves so that the patch is not visible.

SUMMARY:
The most common symptom after an inguinal hernia is postoperative pain. According to the severity of the pain, the quality of life of the patient is also affected. There are many factors associated with postoperative pain. In this study, the results related to the factors affecting postoperative pain were investigated.

DETAILED DESCRIPTION:
The most common symptom after an inguinal hernia is postoperative pain. According to the severity of the pain, the quality of life of the patient is also affected. There are many factors associated with postoperative pain. In the literature, there are factors whose relationship could not be determined clearly in the guidelines prepared for this. A meta-analysis showed that TAPP was associated with less chronic pain than open hernia repair. In another study, it was reported that hernia size and type were unrelated to pain. In the same study, the relationship between preoperative pain and postoperative pain was examined. Etele et al. reported that mesh fixation may increase pain. It is thought that the determination of these multiple predictive factors will both guide postoperative pain management and strengthen patient communication. As a result of the research, it is planned to obtain results related to the factors affecting the postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TAPP for inguinal hernia for the first time

Exclusion Criteria:

* Patients under 18 years of age
* Patients undergoing open hernia repair
* Patients converted from laparoscopic to open
* Patients who are pregnant or likely to become pregnant
* Patients who cannot comply with the treatment or give their own consent for treatment due to their mental state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preoperative demographic data, visual analog scale (VAS) to measure preoperative pain, type and size of inguinal hernia will be evaluated in patients who will undergo TAPP with the diagnosis of inguinal hernia. In the postoperative period, pain intensity will be evaluated on the 1st day, the 3rd day, the 10th day and the 1st month postoperatively. A visual analog scale (VAS) will be applied to the patients for pain scoring. The patients will be followed up for 6 months postoperatively and monitored for complications. The collected data will be statistically analyzed in SPSS.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | one month
  Factors associated with postoperative pain in patients undergoing transabdominal preperitoneal hernia repair due to inguinal hernia will be investigated. A visual analogue scale (VAS) will be used for postoperative pain. Patients will use this scale to score from 0 (no pain) to 10 (worst possible pain) according to their pain status.

CONTACTS AND LOCATIONS:
Overall Officials: Korhan Tuncer, MD, Principal Investigator — Tepecik Training and Research Hospital
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Scheuermann U, Niebisch S, Lyros O, Jansen-Winkeln B, Gockel I. Transabdominal Preperitoneal (TAPP) versus Lichtenstein operation for primary inguinal hernia repair - A systematic review and meta-analysis of randomized controlled trials. BMC Surg. 2017 May 10;17(1):55. doi: 10.1186/s12893-017-0253-7. PMID 28490321
- [Background] Tolver MA, Rosenberg J, Bisgaard T. Early pain after laparoscopic inguinal hernia repair. A qualitative systematic review. Acta Anaesthesiol Scand. 2012 May;56(5):549-57. doi: 10.1111/j.1399-6576.2011.02633.x. Epub 2012 Jan 19. PMID 22260427
- [Background] Etele EE, Neagoe RM, Marton D, Sala D, Torok A. Influence of Mesh Fixation on the Development of Postoperative Pain after Laparoscopic Inguinal Hernia Repair: A Single Surgeon Experience. Chirurgia (Bucur). 2020 Sept-Oct;115(5):609-617. doi: 10.21614/chirurgia.115.5.609. PMID 33138898